CLINICAL TRIAL: NCT00748332
Title: Effects of a Protein-energy Oral Supplement Enriched With Omega-3 Fatty Acids Compared to a Standard Protein-energy Supplement in Cardiac Cachexia
Brief Title: Protein-energy Oral Supplementation Enriched With Omega-3 Fatty Acids in Cardiac Cachexia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: API 2007
Record Dates: First submitted 2008-09-04; First posted 2008-09-08 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2009-06

CONDITIONS: Cardiac Cachexia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Standard oral nutritional supplement
  Interventions: Dietary Supplement: Fortimel Extra®
- 2 (Experimental): Omega-3-enriched oral nutritional supplement
  Interventions: Dietary Supplement: Fortimel Care®

INTERVENTIONS:
Dietary Supplement: Fortimel Extra® — 2 bottles (600 kcal, 40 g proteins) per day
  Arms: 1
Dietary Supplement: Fortimel Care® — Fortimel Care® : 2 bottles (660 kcal, 36 g proteins, 2.38 g EPA) per day
  Arms: 2

SUMMARY:
Cardiac cachexia, the main feature of undernutrition in chronic heart failure, usually defined as a weight loss over 6% over 6 months, is a proven factor of morbidity and mortality in this disease. Its pathophysiology is complex, but proinflammatory cytokines seem to play a major role. Omega-3 poly-unsaturated fatty acids, present in fish oil, have proven beneficial in patients with coronary heart disease, due in part to their effects on membranes but also due to their anti-inflammatory effects, with inhibition of TNF-α and interleukins 1 and 6.

The aim of this phase III randomized controlled double-blinded study is to assess the effects of 8 weeks of a omega-3-enriched protein-energy supplement versus an iso-energetic iso-nitrogenous supplement free of omega-3 fatty acids in cardiac cachexia. Thirty patients will be included in each group. The main judgment criterion will be maximum aerobic capacity (VO2 max), which best reflects aerobic capacity that correlates with muscle mass. Anthropometric, biological (nutritional, inflammatory and involved in food intake control), cardiac (functional) and quality of life will also be studied. All analyses will be performed in intention to treat.

The investigators expect a significantly higher improvement of VO2 max in the omega-3 group.

This study could lead to therapeutic advances in a frequent and severe disease.

DETAILED DESCRIPTION:
Undernutrition is frequent in chronic heart failure (approximately 40%). Cardiac cachexia, main feature of this undernutrition, usually defined as a weight loss over 6% over 6 months, is a proven factor of morbidity and mortality in this disease. Its pathophysiology is complex, but proinflammatory cytokines seem to play a major role, thus appearing close to cancer cachexia. A number of treatments have proven to be effective in preventing undernutrition in chronic heart failure patients (ß-blockers, ACE inhibitors, diuretics and physical training). Omega-3 poly-unsaturated fatty acids, present in fish oil, haven proven beneficial in patients with coronary heart disease, due in part to their effects on membranes but also due to their anti-inflammatory effects, with inhibition of TNF-α and interleukins 1 and 6. However, no study to this day has been conducted in human cardiac cachexia.

The aim of this phase III randomized controlled double-blinded study is to assess the effects of 8 weeks of a omega-3-enriched protein-energy supplement versus an iso-energetic iso-nitrogenous supplement free of omega-3 fatty acids in cardiac cachexia. Thirty patients will be included in each group. The main judgment criterion will be maximum aerobic capacity (VO2 max), which best reflects aerobic capacity that correlates with muscle mass. Anthropometric, biological (nutritional, inflammatory and involved in food intake control), cardiac (functional) and quality of life will also be studied. All analyses will be performed in intention to treat.

We expect a significantly higher improvement of VO2 max in the omega-3 group. This study could lead to therapeutic advances in a frequent and severe disease.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Weight loss between 6 and 10% during the last six months
* Chronic heart failure with end-systolic ejection fraction ≤ 40% (all stages of the NYHA classification)
* Triple therapy: ß-blockers, ACE inhibitors and diuretics
* Informed consent signed
* Affiliated with the French Sécurité Sociale

Exclusion Criteria:

* Patent undernutrition: BMI < 18.5 for ages < 70 or < 21 for ages ≥ 70 and/or weight loss > 10% in the last six months
* Chronic cachectic condition:

  * cancer
  * chronic respiratory failure
  * advanced organ failure
  * hyperthyroidism
  * rheumatoid arthritis
  * AIDS
  * type 1 diabetes
* Drugs affecting muscle mass (e.g., steroids)
* Condition (clinical or EKG) contra-indicating cycle ergometry
* Unstable acute disease
* Edema
* Flare-up of heart failure (BNP > 500 ng/L)
* Intake of omega-3-containing nutritional supplements

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-03; Primary Completion 2011-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
VO2 max (cycle ergometry) | D0 and after 8 weeks

SECONDARY OUTCOMES:
Weight, BMI, body composition (DAX and BIA), muscle function (dynamometers), biology, quality of life, cardiac function (ultra-sound end-systolic ejection fraction, walking perimeter), food intake. | D0 and after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Schneider, PU-PH, Principal Investigator — Department of Gastroentrology of Nice University Hospital
Locations (1):
- Department of Gastro-entérologie, Nice, France